CLINICAL TRIAL: NCT02670915
Title: Efficacy and Safety of Faster-acting Insulin Aspart Compared to NovoRapid® Both in Combination With Insulin Degludec in Children and Adolescents With Type 1 Diabetes
Acronym: onset®7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1218-4101; 2014-002568-33 (EudraCT Number); U1111-1158-1170 (Other: WHO); JapicCTI-163248 (Other: JAPIC)
Record Dates: First submitted 2016-01-27; First posted 2016-02-02 (Estimated); Results first posted 2019-04-04 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-05

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart; insulin degludec

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Meal-time faster-acting insulin aspart and insulin degludec (Experimental)
  Interventions: Drug: Faster-acting insulin aspart; Drug: insulin degludec
- Meal-time NovoRapid® (insulin aspart) and insulin degludec (Active Comparator)
  Interventions: Drug: insulin aspart; Drug: insulin degludec
- Post-meal faster-acting insulin aspart and insulin degludec (Experimental)
  Interventions: Drug: Faster-acting insulin aspart; Drug: insulin degludec

INTERVENTIONS:
Drug: Faster-acting insulin aspart — For subcutaneous (s.c., under the skin) injection once daily.
  Arms: Meal-time faster-acting insulin aspart and insulin degludec; Post-meal faster-acting insulin aspart and insulin degludec
Drug: insulin aspart — For subcutaneous (s.c., under the skin) injection once daily.
  Arms: Meal-time NovoRapid® (insulin aspart) and insulin degludec
Drug: insulin degludec — For subcutaneous (s.c., under the skin) injection once daily.

SUMMARY:
This trial is conducted globally. The aim of the trial is to investigate efficacy and safety of faster-acting insulin aspart compared to NovoRapid® both in combination with insulin degludec in children and adolescents with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria: - Male or female, 1 year above or equal to age below 18 years at the time of signing informed consent and below 18 years at the time of randomisation - Diagnosed with type 1 diabetes mellitus (based on clinical judgement and supported by laboratory analysis as per local guidelines) - Ongoing daily treatment with a basal-bolus insulin regimen using basal insulin analogue or Neutral Protamine Hagedorn (NPH) insulin for at least 90 days prior to the screening visit - HbA1c (glycosylated haemoglobin) below or equal 9.5% (80 mmol/mol) analysed by the central laboratory at the screening visit Exclusion Criteria: - More than one episode of diabetic ketoacidosis requiring hospitalisation within the last 90 days prior to the screening visit - Treatment with any medication for the indication of diabetes or obesity other than stated in the inclusion criteria in a period of 90 days before screening

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 834 (Actual)
Dates: Start 2016-05-04 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (139):
- United States (35):
  - Novo Nordisk Investigational Site, Phoenix, Arizona
  - Novo Nordisk Investigational Site, Tucson, Arizona
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Aurora, Colorado
  - Novo Nordisk Investigational Site, Gainesville, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Tallahassee, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Boise, Idaho
  - Novo Nordisk Investigational Site, Idaho Falls, Idaho
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, Minneapolis, Minnesota
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Neptune City, New Jersey
  - Novo Nordisk Investigational Site, Buffalo, New York
  - Novo Nordisk Investigational Site, Mineola, New York
  - Novo Nordisk Investigational Site, Raleigh, North Carolina
  - Novo Nordisk Investigational Site, Fargo, North Dakota
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Tulsa, Oklahoma
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, Sioux Falls, South Dakota
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
- Bulgaria (3):
  - Novo Nordisk Investigational Site, Pleven
  - Novo Nordisk Investigational Site, Sofia
  - Novo Nordisk Investigational Site, Varna
- Czechia (6):
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Opava
  - Novo Nordisk Investigational Site, Ostrava - Poruba
  - Novo Nordisk Investigational Site, Pardubice
  - Novo Nordisk Investigational Site, Prague
  - Novo Nordisk Investigational Site, Ústí nad Labem
- Estonia (2):
  - Novo Nordisk Investigational Site, Tallinn
  - Novo Nordisk Investigational Site, Tartu
- Finland (3):
  - Novo Nordisk Investigational Site, Espoo
  - Novo Nordisk Investigational Site, OYS
  - Novo Nordisk Investigational Site, Seinäjoki
- Germany (8):
  - Novo Nordisk Investigational Site, Bochum
  - Novo Nordisk Investigational Site, Freiburg im Breisgau
  - Novo Nordisk Investigational Site, Hanover
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Oldenburg
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
- India (9):
  - Novo Nordisk Investigational Site, Hyderabad, Andhra Pradesh
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata
  - Novo Nordisk Investigational Site, New Delhi
- Israel (6):
  - Novo Nordisk Investigational Site, Beersheba
  - Novo Nordisk Investigational Site, Haifa
  - Novo Nordisk Investigational Site, Holon
  - Novo Nordisk Investigational Site, Petah Tikva
  - Novo Nordisk Investigational Site, Tel Aviv
  - Novo Nordisk Investigational Site, Ẕerifin
- Italy (5):
  - Novo Nordisk Investigational Site, Ancona
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Chieti
  - Novo Nordisk Investigational Site, Napoli
  - Novo Nordisk Investigational Site, Verona
- Japan (31):
  - Novo Nordisk Investigational Site, Amagasaki-shi, Hyogo
  - Novo Nordisk Investigational Site, Chuo-shi, Yamanashi
  - Novo Nordisk Investigational Site, Fukuoka
  - Novo Nordisk Investigational Site, Hiroshima-shi, Hiroshima
  - Novo Nordisk Investigational Site, Iruma-gun, Saitama
  - Novo Nordisk Investigational Site, Kitakyushu,Fukuoka
  - Novo Nordisk Investigational Site, Kitakyushu-shi, Fukuoka
  - Novo Nordisk Investigational Site, Kobe-shi, Hyogo
  - Novo Nordisk Investigational Site, Kochi-shi, Kochi
  - Novo Nordisk Investigational Site, Kofu, Yamanashi
  - Novo Nordisk Investigational Site, Kumamoto-shi, Kumamoto
  - Novo Nordisk Investigational Site, Kure-shi, Hiroshima
  - Novo Nordisk Investigational Site, Kyoto
  - Novo Nordisk Investigational Site, Maebashi-shi, Gunma
  - Novo Nordisk Investigational Site, Matsumoto-shi, Nagano,
  - Novo Nordisk Investigational Site, Matsuyama-shi, Ehime
  - Novo Nordisk Investigational Site, Musashino-shi, Tokyo
  - Novo Nordisk Investigational Site, Niigata-shi, Niigata
  - Novo Nordisk Investigational Site, Okayama Kita-ku, Okayama
  - Novo Nordisk Investigational Site, Okayama-shi, Okayama
  - Novo Nordisk Investigational Site, Osaka-shi, Osaka
  - Novo Nordisk Investigational Site, Ota-shi, Gunma
  - Novo Nordisk Investigational Site, Otsu-shi, Shiga
  - Novo Nordisk Investigational Site, Saga-shi, Saga
  - Novo Nordisk Investigational Site, Sendai-shi, Miyagi
  - Novo Nordisk Investigational Site, Suzaka-shi ,Nagano
  - Novo Nordisk Investigational Site, Tochigi
  - Novo Nordisk Investigational Site, Tokyo
  - Novo Nordisk Investigational Site, Tsu-shi, Mie
  - Novo Nordisk Investigational Site, Yokohama-shi, Kanagawa
  - Novo Nordisk Investigational Site, Yokosuka-shi, Kanagawa
- Novo Nordisk Investigational Site, Riga, Latvia
- Novo Nordisk Investigational Site, Kaunas, Lithuania
- Poland (3):
  - Novo Nordisk Investigational Site, Gdansk
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Novo Nordisk Investigational Site, San Juan, Puerto Rico
- Russia (9):
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Novosibirsk
  - Novo Nordisk Investigational Site, Rostov-on-Don
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Samara
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Tomsk
  - Novo Nordisk Investigational Site, Ufa
- Serbia (3):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Novi Sad
- Turkey (Türkiye) (5):
  - Novo Nordisk Investigational Site, Adana
  - Novo Nordisk Investigational Site, Antalya
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Izmir
  - Novo Nordisk Investigational Site, Samsun
- Ukraine (8):
  - Novo Nordisk Investigational Site, Dnipro
  - Novo Nordisk Investigational Site, Ivano-Frankivsk
  - Novo Nordisk Investigational Site, Kharkiv
  - Novo Nordisk Investigational Site, Kiev
  - Novo Nordisk Investigational Site, Kyiv
  - Novo Nordisk Investigational Site, Lviv
  - Novo Nordisk Investigational Site, Vinnytsia
  - Novo Nordisk Investigational Site, Zaporizhzhia

REFERENCES:
- [Background] Bode BW, Iotova V, Kovarenko M, Laffel LM, Rao PV, Deenadayalan S, Ekelund M, Larsen SF, Danne T. Efficacy and Safety of Fast-Acting Insulin Aspart Compared With Insulin Aspart, Both in Combination With Insulin Degludec, in Children and Adolescents With Type 1 Diabetes: The onset 7 Trial. Diabetes Care. 2019 Jul;42(7):1255-1262. doi: 10.2337/dc19-0009. Epub 2019 May 10. PMID 31076415
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 150 sites in 17 countries(number of sites with screened/randomised subjects)-Bulgaria: 4/4; Czech Republic: 6/6; Estonia: 2/2; Finland: 3/3; Germany: 6/6; India: 7/7; Israel: 6/6; Italy: 5/5; Japan: 34/34; Latvia: 1/1; Lithuania: 1/1; Poland: 4/4; Russia: 11/11; Serbia: 4/4; Turkey: 7/7; Ukraine: 9/9; United States: 40/39
Pre-assignment Details: 12-week run-in period: Participants were switched from previous insulin treatment to insulin degludec once daily, and mealtime NovoRapid®/NovoLog®. Insulin degludec treatment was optimised on a weekly basis to the pre-breakfast glycaemic target of 4.0-8.0 mmol/L. Out of 834 participants, who started the run-in period, 57 were run-in failures.
Groups:
- Faster Aspart (Meal): Bolus insulin: Participants received subcutaneous (s.c., into the abdominal wall) injections of faster-acting insulin aspart at mealtime (0-2 minutes before the meal) during the 26-week treatment period. Throughout the trial, the insulin was administered at each of the three main meals (i.e. breakfast, lunch and main evening meal). The insulin was titrated to the pre-meal target of 4.0-8.0 mmol/L, and the bed-time target of 6.7-10 mmol/L in a treat-to-target fashion. Basal insulin: Participants continued insulin degludec once daily s.c. injections from the dose optimization process during the 12-week run-in period till 26-week treatment period. Dose adjustment during the treatment period at the discretion of the investigator was allowed if needed.
- Faster Aspart (Post): Bolus insulin: Participants received s.c. injections of faster-acting insulin aspart at mealtime (20 minutes after the start of the meal) during the 26-week treatment period. Throughout the trial, the insulin was administered at each of the three main meals (i.e. breakfast, lunch and main evening meal). The insulin was titrated to the premeal target of 4.0-8.0 mmol/L, and the bed-time target of 6.7-10 mmol/L in a treat-to-target fashion. Basal insulin: Participants continued insulin degludec once daily s.c. injections from the dose optimization process during the 12-week run-in period till 26-week treatment period. Dose adjustment during the treatment period at the discretion of the investigator was allowed if needed.
- NovoRapid (Meal): Bolus insulin: After 12-week run-in period, participants continued using mealtime insulin aspart (NovoRapid®/NovoLog®) s.c. injections at mealtime (0-2 minutes before the meal) during the 26-week treatment period. Throughout the trial, the insulin was administered at each of the three main meals (i.e. breakfast, lunch and main evening meal). The insulin was titrated to the pre-meal target of 4.0-8.0 mmol/L, and the bed-time target of 6.7-10 mmol/L in a treat-to-target fashion. Basal insulin: Participants continued insulin degludec once daily s.c. injections from the dose optimization process during the 12-week run-in period till 26-week treatment period. Dose adjustment during the treatment period at the discretion of the investigator was allowed if needed.
Period: Overall Study
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Started | 260 | 259 | 258
Completed | 256 | 251 | 253
Not Completed | 4 | 8 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 4
Not completed — Withdrawal by parent/guardian | 4 | 4 | 1
Not completed — Unclassified | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Faster Aspart (Meal): Bolus insulin: Participants received s.c. injections of faster-acting insulin aspart at mealtime (0-2 minutes before the meal) during the 26-week treatment period. Throughout the trial, the insulin was administered at each of the three main meals (i.e. breakfast, lunch and main evening meal). The insulin was titrated to the pre-meal target of 4.0-8.0 mmol/L, and the bed-time target of 6.7-10 mmol/L in a treat-to-target fashion. Basal insulin: Participants continued insulin degludec once daily s.c. injections from the dose optimization process during the 12-week run-in period till 26-week treatment period. Dose adjustment during the treatment period at the discretion of the investigator was allowed if needed.
- Total: Total of all reporting groups
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal) | Total
Number analyzed (Participants) | 260 | 259 | 258 | 777
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.72 (3.74) | 11.62 (3.65) | 11.70 (3.44) | 11.68 (3.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 122 | 110 | 358
  Male | 134 | 137 | 148 | 419
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 17 | 12 | 45
  Not Hispanic or Latino | 244 | 242 | 246 | 732
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 46 | 37 | 43 | 126
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 4 | 5 | 15
  White | 206 | 217 | 209 | 632
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in the Percentage of HbA1c
Description: Change from baseline (week 0) in glycosylated haemoglobin (HbA1c) was evaluated after 26 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In-trial period: the observation period from date of randomisation until last trial-related participant-site contact and included data collected after a subject discontinued trial product.
Time Frame: Week 0, Week 26
Population: Full analysis set (FAS), which included all randomised participants. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Percentage of HbA1c
  Baseline | 7.57 (0.80) | 7.58 (0.84) | 7.53 (0.83)
  Change from baseline: number analyzed (Participants) | 259 | 259 | 258
  Change from baseline | 0.06 (0.80) | 0.33 (0.83) | 0.23 (0.82)
Statistical Analysis 1: Comparison: Faster Aspart (Meal) vs NovoRapid (Meal); The primary analysis was implemented as a statistical model using multiple imputation where the participants without any available HbA1c measurements at scheduled visits had their change from baseline HbA1c value (s) imputed from the available information from the treatment the participant had been randomised to; Test type: Non-Inferiority — Stepwise hierarchical testing procedure was applied: Step 1-Primary analysis: HbA1c non-inferiority of mealtime faster aspart versus mealtime NovoRapid®/NovoLog® both in combination with insulin degludec. Non-inferiority of mealtime faster aspart was considered confirmed if the upper boundary of the two-sided 95% confidence interval (CI) was below or equal to 0.4%; p < 0.001, Multiple imputation — p-values are from the 1-sided test for non-inferiority evaluated at the 2.5% level; Analyses were adjusted for region, strata (age), as factors, and baseline HbA1c as a covariate; Treatment difference = -0.17, 95% CI 2-sided [-0.30 to -0.03]
Statistical Analysis 2: Comparison: Faster Aspart (Post) vs NovoRapid (Meal); The analysis was implemented as a statistical model using multiple imputation where the participants without any available HbA1c measurements at scheduled visits had their change from baseline HbA1c value(s) imputed from the available information from the treatment the participant had been randomised to; Test type: Non-Inferiority — Stepwise hierarchical testing procedure was applied: Step 2-Confirmatory secondary analysis: HbA1c non-inferiority of postmeal faster aspart versus mealtime NovoRapid®/NovoLog® both in combination with insulin degludec. Non-inferiority of mealtime faster aspart was considered confirmed if the upper boundary of the two-sided 95% CI was below or equal to 0.4%; p < 0.001, Multiple imputation — p-values are from the 1-sided test for non-inferiority evaluated at the 2.5% level; Analyses were adjusted for region, strata (age), as factors, and baseline HbA1c as a covariate; Treatment difference = 0.13, 95% CI 2-sided [-0.01 to 0.26]
Statistical Analysis 3: Comparison: Faster Aspart (Meal) vs NovoRapid (Meal); [analysis description as in outcome 1, analysis 2]; Test type: Superiority — Stepwise hierarchical testing procedure was applied: Step 3-Confirmatory secondary analysis: HbA1c superiority of mealtime faster aspart versus mealtime NovoRapid®/NovoLog® both in combination with insulin degludec. Superiority of mealtime faster aspart was considered confirmed if the upper boundary of the two-sided 95% CI was below 0; p = 0.007, multiple imputation — p-values are from the 1-sided test for superiority evaluated at the 2.5% level; Analyses were adjusted for region, strata (age), as factors, and baseline HbA1c as a covariate; Treatment difference = -0.17, 95% CI 2-sided [-0.30 to -0.03]

2. Secondary Outcome: Change in 8-point SMPG Profile: Mean PPG Over All Three Meals
Description: Change from baseline (week 0) in mean post prandial glucose (PPG) over all three meals was evaluated after 26 weeks of randomisation. PPG for each meal (breakfast, lunch and main evening meal) was recorded by the participant as part of the 8-point self-measured plasma glucose (SMPG) profile. Mean PPG over all three meals was derived as the mean of all corresponding mean meal. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 210 | 221 | 214
  Baseline | 10.19 (2.64) | 10.12 (2.79) | 10.03 (2.52)
  Change from baseline: number analyzed (Participants) | 196 | 200 | 203
  Change from baseline | -0.94 (2.55) | 0.36 (3.17) | -0.21 (2.79)

3. Secondary Outcome: Change in 8-point SMPG Profile: PPG Increment Over All Three Meals
Description: Change from baseline (week 0) in mean PPG increment over all three meals was evaluated after 26 weeks of randomisation. Postprandial glucose (PPG) increment for each meal (breakfast, lunch and main evening meal) was derived from the 8-point profile as the difference between PPG (1 hour after the meal) values and the plasma glucose (PG) value before meal. The mean of the derived increments was then calculated separately for each meal. Mean PPG increment over all three meals was derived as the mean of all corresponding mean meal increments. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis. .
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 210 | 219 | 213
  Baseline | 1.20 (2.70) | 1.01 (2.48) | 0.97 (2.55)
  Change from baseline: number analyzed (Participants) | 196 | 197 | 202
  Change from baseline | -0.92 (2.92) | 0.56 (2.88) | 0.14 (2.75)

4. Secondary Outcome: Change in 8-point SMPG Profile: Individual Meal (Breakfast, Lunch and Main Evening Meal) PPG
Description: Change from baseline (week 0) in individual meal (breakfast, lunch and main evening meal) PPG was evaluated after 26 weeks of randomisation. PPG for each meal was recorded by the participant as part of the 8-point SMPG profile. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Breakfast: Baseline: number analyzed (Participants) | 227 | 235 | 236
  Breakfast: Baseline | 10.51 (3.59) | 10.51 (3.77) | 10.49 (3.59)
  Breakfast: Change from baseline: number analyzed (Participants) | 216 | 217 | 229
  Breakfast: Change from baseline | -1.11 (3.91) | 0.16 (3.95) | 0.04 (3.89)
  Lunch: Baseline: number analyzed (Participants) | 227 | 232 | 229
  Lunch: Baseline | 9.69 (3.32) | 9.99 (3.82) | 9.62 (3.30)
  Lunch: Change from baseline: number analyzed (Participants) | 215 | 220 | 223
  Lunch: Change from baseline | -0.80 (3.74) | 0.18 (4.40) | -0.24 (4.22)
  Main evening meal: Baseline: number analyzed (Participants) | 228 | 231 | 231
  Main evening meal: Baseline | 10.24 (3.64) | 9.90 (3.59) | 9.87 (3.46)
  Main evening meal: Change from baseline: number analyzed (Participants) | 222 | 220 | 225
  Main evening meal: Change from baseline | -0.74 (3.96) | 0.61 (4.40) | -0.05 (4.14)

5. Secondary Outcome: Change in 8-point SMPG Profile: Individual Meal (Breakfast, Lunch and Main Evening Meal) PPG Increment
Description: Change from baseline (week 0) in individual meal (breakfast, lunch and main evening meal) PPG increment was evaluated after 26 weeks of randomisation. PPG increment for each meal was derived from the 8-point profile as the difference between PPG values (1 hour after the meal) and the PG value before meal. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Breakfast: Baseline: number analyzed (Participants) | 227 | 235 | 235
  Breakfast: Baseline | 1.90 (3.64) | 2.10 (3.59) | 2.12 (4.08)
  Breakfast: Change from baseline: number analyzed (Participants) | 216 | 217 | 228
  Breakfast: Change from baseline | -0.82 (4.44) | 0.46 (4.21) | 0.10 (4.66)
  Lunch: Baseline: number analyzed (Participants) | 227 | 231 | 229
  Lunch: Baseline | 1.02 (3.82) | 1.12 (3.79) | 0.74 (3.88)
  Lunch: Change from baseline: number analyzed (Participants) | 215 | 219 | 222
  Lunch: Change from baseline | -0.58 (4.92) | 0.12 (4.41) | -0.11 (4.54)
  Main evening meal: Baseline: number analyzed (Participants) | 228 | 230 | 231
  Main evening meal: Baseline | 0.53 (4.28) | -0.26 (3.53) | -0.06 (3.78)
  Main evening meal: Change from baseline: number analyzed (Participants) | 222 | 218 | 225
  Main evening meal: Change from baseline | -0.92 (5.07) | 1.03 (4.68) | 0.45 (4.31)

6. Secondary Outcome: Change in 8-point SMPG Profile: Mean of the 8-point Profile
Description: Change from baseline (week 0) in mean of the 8-point SMPG profile was evaluated after 26 weeks of randomisation. SMPG values were recorded at 8 time-points on two consecutive days: before and after (60 minute after the start of the meal) breakfast, lunch and main evening meal, before bedtime, and before breakfast on the next day. Mean of the 8-point profile was derived as the mean of all corresponding mean SMPG recorded at 8 different time points. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 240 | 242 | 246
  Baseline | 9.41 (1.98) | 9.47 (1.89) | 9.39 (1.97)
  Change from baseline: number analyzed (Participants) | 235 | 235 | 245
  Change from baseline | -0.27 (2.04) | 0.17 (2.12) | -0.05 (2.29)

7. Secondary Outcome: Fluctuation in the 8-point SMPG Profile
Description: Fluctuation in the 8-point SMPG profile was evaluated after 26 weeks of randomisation. Fluctuation in 8-point SMPG profile was the average absolute difference from the mean of the SMPG profile. The results are based on the last in-trial value.
Time Frame: Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L | 1.88 (44.49) | 1.94 (42.51) | 1.83 (45.98)

8. Secondary Outcome: Change in FPG
Description: Change from baseline (week 0) in fasting plasma glucose (FPG) was evaluated after 26 weeks of randomisation. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 186 | 198 | 180
  Baseline | 7.58 (3.56) | 8.03 (3.35) | 7.79 (3.48)
  Change from baseline: number analyzed (Participants) | 173 | 185 | 161
  Change from baseline | 0.41 (5.04) | -0.08 (4.49) | -0.13 (4.16)

9. Secondary Outcome: Change in 1,5-anhydroglucitol
Description: Change from baseline (week 0) in 1,5-anhydroglucitol was evaluated after 26 weeks of randomisation. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
ug/mL
  Baseline: number analyzed (Participants) | 258 | 257 | 254
  Baseline | 4.95 (3.62) | 5.07 (3.97) | 5.13 (3.76)
  Change from baseline: number analyzed (Participants) | 257 | 257 | 254
  Change from baseline | -0.06 (3.13) | -0.85 (2.80) | -0.63 (2.42)

10. Secondary Outcome: Percentage of Subjects Reaching HbA1c Target (HbA1c Less Than 7.5 %) According to ISPAD Guidelines
Description: Percentage of participants (yes/no) reaching HbA1c less than 7.5 % according to International Society for Pediatric and Adolescent Diabetes (ISPAD) guidelines was evaluated after 26 weeks of randomisation. The results are based on the last in-trial value.
Time Frame: Week 26
Population: FAS.
Measure: Number; unit: Percentage of participants
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Percentage of participants
  Yes | 42.3 | 31.7 | 39.5
  No | 57.7 | 68.3 | 60.5

11. Secondary Outcome: Percentage of Subjects Reaching HbA1c Target (HbA1c Less Than 7.5 %) According to ISPAD Guidelines, Without Severe Hypoglycaemia
Description: Percentage of participants (yes/no) reaching HbA1c less than 7.5 % according to ISPAD guidelines, without severe hypoglycaemia was evaluated after 26 weeks of randomisation. Severe hypoglycaemia according to ISPAD guidelines: hypoglycaemic episode associated with severe neuroglycopenia, usually resulting in coma or seizure and requiring parenteral therapy (glucagon or intravenous glucose). The results are based on the last in-trial value.
Time Frame: Week 26
Population: FAS.
Measure: Number; unit: Percentage of participants
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Percentage of participants
  Yes | 41.9 | 30.9 | 38.4
  No | 58.1 | 69.1 | 61.6

12. Secondary Outcome: Insulin Dose (Units/Day): Total Basal
Description: Total basal insulin dose (Units/day) was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period: the observation period from date of first dose of randomised NovoRapid®/NovoLog® / faster aspart and no later than 7 days after the day of last dose of NovoRapid®/NovoLog® / faster aspart. The on-treatment observation period includes data collected up to and including 7 days after treatment discontinuation. Number of participants analysed = number of participants contributed to the analysis. Analysis population description: Safety analysis set (SAS) included all participants receiving at least one dose of the investigational product (faster aspart) or its comparator (NovoRapid®/NovoLog®).
Time Frame: Week 26
Population: SAS. One participant was randomised to the postmeal faster aspart group but was exposed to mealtime faster aspart throughout the study. The participant was included in the mealtime faster aspart group for the SAS. Therefore, number of participants analysed = Faster aspart (meal): 261, Faster aspart (post): 258 and NovoRapid (meal): 258.
Measure: Mean (Standard Deviation); unit: Units (U)
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Units (U) | 21.6 (12.9) | 21.5 (14.5) | 20.7 (12.8)

13. Secondary Outcome: Insulin Dose (Units/Day): Total Bolus
Description: Total bolus insulin dose (Units/day) was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 26
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units (U)
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Units (U) | 23.3 (14.5) | 23.5 (15.1) | 22.5 (13.0)

14. Secondary Outcome: Insulin Dose (Units/Day): Individual Meal Insulin Dose
Description: Individual meal (breakfast, lunch and main evening meal) insulin dose (Units/day) was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value.
Time Frame: Week 26
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units (U)
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Units (U)
  Breakfast | 7.3 (5.1) | 7.1 (4.9) | 6.8 (4.4)
  Lunch | 8.1 (5.1) | 8.4 (6.2) | 7.9 (5.2)
  Main evening meal | 8.1 (6.0) | 8.0 (5.4) | 7.7 (5.1)

15. Secondary Outcome: Insulin Dose (Units/kg/Day): Total Basal
Description: Total basal insulin dose (Units/kg/day) was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 26
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units (U)/kg
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Units (U)/kg | 0.433 (0.228) | 0.425 (0.196) | 0.409 (0.176)

16. Secondary Outcome: Insulin Dose (Units/kg/Day): Total Bolus
Description: Total bolus insulin dose (Units/kg/day) was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 26
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units (U)/kg
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Units (U)/kg | 0.483 (0.256) | 0.491 (0.241) | 0.468 (0.224)

17. Secondary Outcome: Insulin Dose (Units/kg/Day): Individual Meal Insulin Dose
Description: Individual meal (breakfast, lunch and main evening meal) insulin dose (Units/kg/day) was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 26
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units (U)/kg
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Units (U)/kg
  Breakfast | 0.151 (0.091) | 0.150 (0.079) | 0.144 (0.081)
  Lunch | 0.170 (0.103) | 0.174 (0.104) | 0.166 (0.095)
  Main evening meal | 0.164 (0.099) | 0.165 (0.092) | 0.158 (0.086)

18. Secondary Outcome: Change of Time Spent in Low Interstitial Glucose (IG) (IG <=3.9 mmol/L [70 mg/dL])
Description: Change from baseline (week 0) in the time spent in low IG (<=3.9 mmol/L [70 mg/dL]) based on continuous glucose monitoring (CGM) was evaluated after 26 weeks of randomisation. A subgroup of participants wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Minutes/day
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Minutes/day
  Baseline: number analyzed (Participants) | 43 | 48 | 44
  Baseline | 107.94 (77.34) | 100.70 (77.28) | 81.52 (71.90)
  Change from baseline: number analyzed (Participants) | 42 | 46 | 41
  Change from baseline | -24.11 (71.74) | -13.06 (82.55) | 6.92 (74.64)

19. Secondary Outcome: Incidence of Episodes With IG <=2.5, 3.0, 3.9 mmol/L (45, 54, 70 mg/dL) and IG >10.0, 12.0 mmol/L (180, 216 mg/dL)
Description: Incidence of episodes (number of episodes per 24 hours) with IG <=2.5, 3.0, 3.9 mmol/L (45, 54, 70 mg/dL) and IG >10.0, 12.0 mmol/L (180, 216 mg/dL) based on CGM was calculated after 26 weeks of randomisation. A subgroup of participants wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. The results are based on the last in-trial value.
Time Frame: Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Number; unit: Episodes per 24 hours
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes per 24 hours
  Episodes with IG <=2.5 mmol/L: number analyzed (Participants) | 36 | 36 | 32
  Episodes with IG <=2.5 mmol/L | 0.55 | 0.68 | 0.57
  Episodes with IG <=3.0 mmol/L: number analyzed (Participants) | 39 | 42 | 36
  Episodes with IG <=3.0 mmol/L | 1.01 | 1.10 | 1.03
  Episodes with IG <=3.9 mmol/L: number analyzed (Participants) | 42 | 45 | 39
  Episodes with IG <=3.9 mmol/L | 2.29 | 2.30 | 2.24
  Episodes with IG >10 mmol/L: number analyzed (Participants) | 42 | 46 | 41
  Episodes with IG >10 mmol/L | 11.52 | 11.61 | 11.65
  Episodes with IG >12 mmol/L: number analyzed (Participants) | 42 | 46 | 41
  Episodes with IG >12 mmol/L | 7.64 | 7.77 | 8.05

20. Secondary Outcome: Percentage of Time Spent With IG <=2.5, 3.0, 3.9 mmol/L (45, 54, 70 mg/dL) and IG >10.0, 12.0 mmol/L (180, 216 mg/dL)
Description: Percentage of time spent with IG <=2.5, 3.0, 3.9 mmol/L (45, 54, 70 mg/dL) and IG >10.0, 12.0 mmol/L (180, 216 mg/dL) based on CGM was evaluated after 26 weeks of randomisation. A subgroup of participants wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. The results are based on the last in-trial value.
Time Frame: Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Percentage of time
  Time spent with IG <=2.5 mmol/L: number analyzed (Participants) | 42 | 46 | 41
  Time spent with IG <=2.5 mmol/L | 1.09 (1.50) | 1.80 (3.21) | 1.34 (1.90)
  Time spent with IG <=3.0 mmol/L: number analyzed (Participants) | 42 | 46 | 41
  Time spent with IG <=3.0 mmol/L | 2.19 (2.35) | 2.90 (4.06) | 2.48 (2.92)
  Time spent with IG <=3.9 mmol/L: number analyzed (Participants) | 42 | 46 | 41
  Time spent with IG <=3.9 mmol/L | 5.97 (4.59) | 6.25 (5.68) | 5.97 (5.38)
  Time spent with IG >10 mmol/L: number analyzed (Participants) | 42 | 46 | 41
  Time spent with IG >10 mmol/L | 40.40 (14.80) | 40.60 (14.38) | 42.47 (17.51)
  Time spent with IG >12 mmol/L: number analyzed (Participants) | 42 | 46 | 41
  Time spent with IG >12 mmol/L | 26.09 (12.82) | 25.67 (13.60) | 28.62 (16.83)

21. Secondary Outcome: Percentage of Time Spent Within IG Target 4.0-10.0 mmol/L (71-180 mg/dL) Both Included
Description: Percentage of time spent within IG target 4.0-10.0 mmol/L (71-180 mg/dL), both included based on CGM was evaluated after 26 weeks of randomisation. A subgroup of participants wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. The results are based on the last in-trial value.
Time Frame: Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of time
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Percentage of time | 53.00 (12.15) | 52.56 (14.08) | 51.03 (16.25)

22. Secondary Outcome: Change in Mean IG Increment (0-1 Hours and 0-2 Hours After Start of the Meal)
Description: Change from baseline (week 0) in mean IG increment (0-1 hours and 0-2 hours after start of the meal) based on CGM was evaluated after 26 weeks of randomisation. A subgroup of participants wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. Presented values are mean of all the meals (breakfast, lunch and evening meal). The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  0-1 hour: Baseline: number analyzed (Participants) | 37 | 45 | 41
  0-1 hour: Baseline | 0.56 (0.58) | 0.73 (0.54) | 0.61 (0.49)
  0-1 hour: Change from baseline: number analyzed (Participants) | 36 | 41 | 40
  0-1 hour: Change from baseline | -0.19 (0.55) | 0.26 (0.83) | 0.07 (0.50)
  0-2 hour: Baseline: number analyzed (Participants) | 37 | 45 | 41
  0-2 hour: Baseline | 0.76 (0.75) | 1.10 (1.03) | 0.86 (0.69)
  0-2 hour: Change from baseline: number analyzed (Participants) | 36 | 41 | 40
  0-2 hour: Change from baseline | -0.35 (0.87) | 0.55 (1.14) | 0.09 (0.59)

23. Secondary Outcome: Change in Mean IG Peak After Start of Meal
Description: Change from baseline (week 0) in mean IG peak after start of meal based on CGM was evaluated after 26 weeks of randomisation. A subgroup of participants wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. Presented values are mean of all the meals (breakfast, lunch and evening meal). The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 37 | 45 | 41
  Baseline | 12.90 (1.88) | 12.92 (1.97) | 12.90 (2.25)
  Change from baseline: number analyzed (Participants) | 37 | 42 | 40
  Change from baseline | -0.28 (1.91) | 0.80 (1.84) | 0.38 (2.00)

24. Secondary Outcome: Change in Mean Time to the IG Peak After Meal
Description: Change from baseline (week 0) in mean time to the IG peak after meal based on CGM was evaluated after 26 weeks of randomisation. A subgroup of subjects wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. Presented values are mean of all the meals (breakfast, lunch and evening meal). The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Minutes
  Baseline: number analyzed (Participants) | 37 | 45 | 41
  Baseline | 103.16 (16.87) | 106.21 (20.68) | 102.20 (17.09)
  Change from baseline: number analyzed (Participants) | 37 | 42 | 40
  Change from baseline | 4.70 (25.85) | -8.56 (22.62) | 2.29 (19.80)

25. Secondary Outcome: Change in 30-minute PPG
Description: Change from baseline (week 0) in 30-minute PPG based on meal test was evaluated after 26 weeks of randomisation. In connection to wearing the CGM for 11 to 13 days up to week 0 and up to week 26, the subgroup of participants had a standardised liquid meal test at the 2 visits, monitoring the PPG at 30-minute after the meal intake at the visit. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 41 | 46 | 40
  Baseline | 11.28 (3.26) | 10.96 (3.78) | 11.71 (3.13)
  Change from baseline: number analyzed (Participants) | 40 | 45 | 39
  Change from baseline | -0.21 (3.49) | 1.84 (3.41) | -0.45 (3.42)

26. Secondary Outcome: Change in 30-minute PPG Increment
Description: Change from baseline (week 0) in 30-minute PPG increment based on meal test was evaluated after 26 weeks of randomisation. In connection to wearing the CGM for 11 to 13 days up to week 0 and up to week 26, the subgroup of participants had a standardised liquid meal test at the 2 visits, monitoring the pre-prandial glucose (before the meal) the PPG at 30-minute (after the meal) at the visit. PPG increment was derived as 30-minute PPG measurement minus the pre-prandial PG. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 41 | 46 | 40
  Baseline | 3.44 (2.16) | 3.48 (2.50) | 4.02 (2.18)
  Change from baseline: number analyzed (Participants) | 40 | 44 | 39
  Change from baseline | 0.36 (2.92) | 1.92 (2.79) | -0.34 (2.18)

27. Secondary Outcome: Change in 1-hour PPG
Description: Change from baseline (week 0) in 1-hour PPG based on meal test was evaluated after 26 weeks of randomisation. In connection to wearing the CGM for 11 to 13 days up to week 0 and up to week 26, the subgroup of participants had a standardised liquid meal test at the 2 visits, monitoring the PPG at 1-hour after the meal intake at the visit. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 41 | 46 | 40
  Baseline | 12.77 (3.92) | 12.56 (5.08) | 13.06 (3.86)
  Change from baseline: number analyzed (Participants) | 40 | 45 | 39
  Change from baseline | -0.15 (4.39) | 2.54 (4.43) | -0.63 (4.73)

28. Secondary Outcome: Change in 1-hour PPG Increment
Description: Change from baseline (week 0) in 1-hour PPG increment based on meal test was evaluated after 26 weeks of randomisation. In connection to wearing the CGM for 11 to 13 days up to week 0 and up to week 26, the subgroup of participants had a standardised liquid meal test at the 2 visits, monitoring the pre-prandial glucose (before the meal) the PPG at 1-hour (after the meal) at the visit. PPG increment was derived as 1-hour PPG measurement minus the pre-prandial PG. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 41 | 46 | 40
  Baseline | 4.93 (3.34) | 5.08 (4.21) | 5.36 (2.77)
  Change from baseline: number analyzed (Participants) | 40 | 44 | 39
  Change from baseline | 0.42 (4.93) | 2.63 (4.03) | -0.52 (3.17)

29. Secondary Outcome: Change in 2-hour PPG
Description: Change from baseline (week 0) in 2-hour PPG based on meal test was evaluated after 26 weeks of randomisation. In connection to wearing the CGM for 11 to 13 days up to week 0 and up to week 26, the subgroup of participants had a standardised liquid meal test at the 2 visits, monitoring the PPG at 2-hour after the meal intake at the visit. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 41 | 46 | 40
  Baseline | 12.50 (4.63) | 12.54 (5.74) | 12.37 (4.74)
  Change from baseline: number analyzed (Participants) | 40 | 45 | 39
  Change from baseline | 0.69 (5.88) | 1.80 (5.08) | -0.75 (5.64)

30. Secondary Outcome: Change in 2-hour PPG Increment
Description: Change from baseline (week 0) in 2-hour PPG increment based on meal test was evaluated after 26 weeks of randomisation. In connection to wearing the CGM for 11 to 13 days up to week 0 and up to week 26, the subgroup of participants had a standardised liquid meal test at the 2 visits, monitoring the pre-prandial glucose (before the meal) the PPG at 2-hour (after the meal) at the visit. PPG increment was derived as 2-hour PPG measurement minus the pre-prandial PG. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 41 | 46 | 40
  Baseline | 4.66 (4.22) | 5.06 (5.04) | 4.67 (3.83)
  Change from baseline: number analyzed (Participants) | 40 | 44 | 39
  Change from baseline | 1.26 (6.81) | 1.62 (5.03) | -0.64 (4.43)

31. Secondary Outcome: Change in AUCIG,0-15min
Description: Change in area under the IG curve 0-15 minutes post meal (AUCIG,0-15min) during meal test and based on CGM measurements was evaluated after 26 weeks of randomisation. Interstitial glucose (IG) was measured every 5 minutes. The endpoint was calculated as the area under the IG curve using the trapezoidal method and weighted by duration. A subgroup of participants wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 37 | 43 | 40
  Baseline | 8.01 (2.72) | 7.49 (2.07) | 7.66 (1.96)
  Change from baseline: number analyzed (Participants) | 34 | 41 | 38
  Change from baseline | -1.27 (3.68) | 0.08 (2.48) | -0.53 (2.85)

32. Secondary Outcome: Change in AUCIG,0-30min
Description: Change in area under the IG curve 0-30 minutes post meal (AUCIG,0-30min) during meal test and based on CGM measurements was evaluated after 26 weeks of randomisation. IG was measured every 5 minutes. The endpoint was calculated as the area under the IG curve using the trapezoidal method and weighted by duration. A subgroup of participants wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 37 | 43 | 40
  Baseline | 8.28 (2.75) | 7.80 (2.13) | 8.13 (1.87)
  Change from baseline: number analyzed (Participants) | 34 | 41 | 38
  Change from baseline | -1.15 (3.62) | 0.22 (2.52) | -0.47 (2.81)

33. Secondary Outcome: Change in AUCIG,0-1h
Description: Change in area under the IG curve 0-1 hour post meal (AUCIG,0-1h) during meal test and based on CGM measurements was evaluated after 26 weeks of randomisation. IG was measured every 5 minutes. The endpoint was calculated as the area under the IG curve using the trapezoidal method and weighted by duration. A subgroup of participants wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 37 | 44 | 40
  Baseline | 9.63 (2.90) | 9.43 (2.71) | 10.02 (2.19)
  Change from baseline: number analyzed (Participants) | 34 | 42 | 38
  Change from baseline | -0.87 (3.71) | 0.54 (3.00) | -0.65 (2.91)

34. Secondary Outcome: Change in AUCIG,0-2h
Description: Change in area under the IG curve 0-2 hours post meal (AUCIG,0-2h) during meal test and based on CGM measurements was evaluated after 26 weeks of randomisation. IG was measured every 5 minutes. The endpoint was calculated as the area under the IG curve using the trapezoidal method and weighted by duration. A subgroup of participants wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 38 | 44 | 40
  Baseline | 11.40 (3.20) | 11.48 (3.43) | 11.76 (2.80)
  Change from baseline: number analyzed (Participants) | 35 | 42 | 38
  Change from baseline | -0.84 (3.93) | 0.75 (3.74) | -0.86 (3.61)

35. Secondary Outcome: Change in AUCIG,0-4h
Description: Change in area under the IG curve 0-4 hours post meal (AUCIG,0-4h) during meal test and based on CGM measurements was evaluated after 26 weeks of randomisation. IG was measured every 5 minutes. The endpoint was calculated as the area under the IG curve using the trapezoidal method and weighted by duration. A subgroup of participants wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 38 | 44 | 40
  Baseline | 11.21 (3.25) | 11.19 (3.47) | 11.46 (3.21)
  Change from baseline: number analyzed (Participants) | 35 | 42 | 38
  Change from baseline | -0.38 (3.96) | 0.62 (3.97) | -1.30 (4.13)

36. Secondary Outcome: Change in Time to the IG Peak After Start of Meal
Description: Change in time to the IG peak after start of meal during meal test and based on CGM measurements was evaluated after 26 weeks of randomisation. A subgroup of participants wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. Presented values are mean of all the meals (breakfast, lunch and evening meal). The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Minute
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Minute
  Baseline: number analyzed (Participants) | 38 | 44 | 40
  Baseline | 102.85 (48.93) | 94.26 (38.22) | 93.80 (39.19)
  Change from baseline: number analyzed (Participants) | 35 | 42 | 38
  Change from baseline | 5.29 (55.42) | -0.04 (42.05) | -8.76 (52.17)

37. Secondary Outcome: Change in IG Peak After Start of Meal
Description: Change in IG peak after start of meal during meal test and based on CGM measurements was evaluated after 26 weeks of randomisation. A subgroup of participants wore a CGM for between 11 and 13 days up to week 0 (randomisation) and up to week 26 to monitor their IG on a continuous basis. Presented values are mean of all the meals (breakfast, lunch and evening meal). The results are based on the last in-trial value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline: number analyzed (Participants) | 38 | 44 | 40
  Baseline | 14.87 (3.55) | 15.15 (4.52) | 15.11 (3.62)
  Change from baseline: number analyzed (Participants) | 35 | 42 | 38
  Change from baseline | -0.55 (3.77) | 1.11 (4.88) | -1.36 (4.36)

38. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to American Diabetes Association (ADA)/ISPAD Classification: Total
Description: Treatment emergent: if the onset of the episode occurred on or after the first day of treatment with investigational medicinal product (IMP) after randomisation, and no later than 1 day after the last day on IMP. Classification of hypoglycaemia: 1) Severe (according to ISPAD classification). Following are according to ADA classification: 2) Documented symptomatic: episode during which typical symptoms of hypoglycaemia are accompanied by a PG level ≤3.9 mmol/L. 3) Asymptomatic: episode not accompanied by typical symptoms of hypoglycaemia, but with a PG level ≤3.9 mmol/L. 4) Probable symptomatic: an episode during which symptoms of hypoglycaemia are not accompanied by a PG determination but that was presumably caused by a PG level ≤3.9 mmol/L. 5) Pseudo-hypoglycaemia: episode during which the person with diabetes reports any of the typical symptoms of hypoglycaemia with a PG level >3.9mmol/L, but approaching that level. The results are based on the on-treatment period.
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 3 | 8 | 4
  Documented symptomatic | 5391 | 5712 | 5170
  Asymptomatic | 4255 | 3781 | 3656
  Probable symptomatic | 12 | 10 | 24
  Pseudo-hypoglycaemia | 35 | 37 | 47
  Unclassifiable | 5 | 2 | 1

39. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to ADA/ISPAD Classification: Daytime
Description: Classification of hypoglycaemia: 1) Severe (according to ISPAD classification). Following are according to ADA classification: 2) Documented symptomatic. 3) Asymptomatic. 4) Probable symptomatic. 5) Pseudo-hypoglycaemia. Daytime period: The period between 07:01 and 22:59 (both included). The results are based on the on-treatment period.
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 3 | 5 | 3
  Documented symptomatic | 4895 | 5077 | 4779
  Asymptomatic | 3584 | 3163 | 3101
  Probable symptomatic | 10 | 10 | 22
  Pseudo-hypoglycaemia | 32 | 31 | 42
  Unclassifiable | 5 | 2 | 1

40. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to ADA/ISPAD Classification: Nocturnal (23:00-7:00, Both Included)
Description: Classification of hypoglycaemia: 1) Severe (according to ISPAD classification). Following are according to ADA classification: 2) Documented symptomatic. 3) Asymptomatic. 4) Probable symptomatic. 5) Pseudo-hypoglycaemia. Nocturnal period: The period between 23:00 and 07:00 (both included). The results are based on the on-treatment period.
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 0 | 3 | 1
  Documented symptomatic | 496 | 635 | 391
  Asymptomatic | 671 | 618 | 555
  Probable symptomatic | 2 | 0 | 2
  Pseudo-hypoglycaemia | 3 | 6 | 5
  Unclassifiable | 0 | 0 | 0

41. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to Novo Nordisk/ISPAD Classification: Total
Description: Classification of hypoglycaemia: 1) Severe (according to ISPAD classification). Following are according to Novo Nordisk classification: 2) Symptomatic blood glucose (BG) confirmed: episode that is BG confirmed by PG value <3.1 mmol/L (56 mg/dL) with symptoms consistent with hypoglycaemia. 3) Asymptomatic BG confirmed: episode that is BG confirmed by PG value <3.1 mmol/L without symptoms consistent with hypoglycaemia. 4) Severe or BG confirmed symptomatic: an episode that is severe according to the ISPAD classification or BG confirmed by a PG value <3.1 mmol/L with symptoms consistent with hypoglycaemia. 5) BG confirmed: an episode that is BG confirmed by a PG value <3.1 mmol/L with or without symptoms consistent with hypoglycaemia. 6) Severe or BG confirmed: an episode that is severe according to the ISPAD Classification or BG confirmed by a PG value <3.1 mmol/L with or without symptoms consistent with hypoglycaemia. The results are based on the on-treatment period.
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 3 | 8 | 4
  BG confirmed | 3580 | 3586 | 3272
  Severe or BG confirmed symptomatic | 2242 | 2427 | 2194
  Severe or BG confirmed | 3583 | 3594 | 3276
  Unclassifiable | 6118 | 5956 | 5626

42. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to Novo Nordisk/ISPAD Classification: Daytime
Description: Classification of hypoglycaemia: 1) Severe (according to ISPAD classification). Following are according to Novo Nordisk classification: 2) BG confirmed. 3) Severe or BG confirmed symptomatic. 4) Severe or BG confirmed. 5) Asymptomatic BG confirmed. Daytime period: The period between 07:01 and 22:59 (both included). The results are based on the on-treatment period.
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 3 | 5 | 3
  BG confirmed | 3184 | 3112 | 2960
  Severe or BG confirmed symptomatic | 2062 | 2167 | 2035
  Severe or BG confirmed | 3187 | 3117 | 2963
  Unclassifiable | 5342 | 5171 | 4985

43. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to Novo Nordisk/ISPAD Classification: Nocturnal (23:00-7:00, Both Included)
Description: Classification of hypoglycaemia: 1) Severe (according to ISPAD classification). Following are according to Novo Nordisk classification: 2) BG confirmed. 3) Severe or BG confirmed symptomatic. 4) Severe or BG confirmed. 5) Asymptomatic BG confirmed. Nocturnal period: The period between 23:00 and 07:00 (both included). The results are based on the on-treatment period.
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 0 | 3 | 1
  BG confirmed | 396 | 474 | 312
  Severe or BG confirmed symptomatic | 180 | 260 | 159
  Severe or BG confirmed | 396 | 477 | 313
  Unclassifiable | 776 | 785 | 641

44. Secondary Outcome: Number of Treatment Emergent Meal Related (From Start of Meal Until 1 Hour After Start of Meal) Hypoglycaemic Episodes According to ADA/ISPAD Classification
Description: Classification of hypoglycaemia: 1) Severe (according to ISPAD classification). Following are according to ADA classification: 2) Documented symptomatic. 3) Asymptomatic. 4) Probable symptomatic. 5) Pseudo-hypoglycaemia. The results are based on the on-treatment period.
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 0 | 0 | 0
  Documented symptomatic | 178 | 113 | 157
  Asymptomatic | 77 | 51 | 55
  Probable symptomatic | 0 | 0 | 1
  Pseudo-hypoglycaemia | 1 | 2 | 1
  Unclassifiable | 0 | 0 | 0

45. Secondary Outcome: Number of Treatment Emergent Meal Related (From Start of Meal Until 2 Hours After Start of Meal) Hypoglycaemic Episodes According to ADA/ISPAD Classification
Description: as for outcome 44
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 2 | 1 | 1
  Documented symptomatic | 1125 | 882 | 1016
  Asymptomatic | 421 | 268 | 303
  Probable symptomatic | 1 | 1 | 7
  Pseudo-hypoglycaemia | 6 | 6 | 4
  Unclassifiable | 0 | 0 | 0

46. Secondary Outcome: Number of Treatment Emergent Meal Related (From Start of Meal Until 4 Hours After Start of Meal) Hypoglycaemic Episodes According to ADA/ISPAD Classification
Description: as for outcome 44
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 3 | 1 | 2
  Documented symptomatic | 3041 | 3064 | 2812
  Asymptomatic | 1340 | 1194 | 1168
  Probable symptomatic | 4 | 8 | 16
  Pseudo-hypoglycaemia | 15 | 18 | 17
  Unclassifiable | 2 | 0 | 0

47. Secondary Outcome: Number of Treatment Emergent Meal Related (From 2-4 Hours After Start of Meal) Hypoglycaemic Episodes According to ADA/ISPAD Classification
Description: as for outcome 44
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 1 | 0 | 1
  Documented symptomatic | 1916 | 2182 | 1796
  Asymptomatic | 919 | 926 | 865
  Probable symptomatic | 3 | 7 | 9
  Pseudo-hypoglycaemia | 9 | 12 | 13
  Unclassifiable | 2 | 0 | 0

48. Secondary Outcome: Number of Treatment Emergent Meal Related (From Start of Meal Until 1 Hour After Start of Meal) Hypoglycaemic Episodes According to Novo Nordisk/ISPAD Classification
Description: Classification of hypoglycaemia: 1) Severe (according to ISPAD classification). Following are according to Novo Nordisk classification: 2) BG confirmed. 3) Severe or BG confirmed symptomatic. 4) Severe or BG confirmed. 5) Asymptomatic BG confirmed. The results are based on the on-treatment period.
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 0 | 0 | 0
  BG confirmed | 119 | 66 | 105
  Severe or BG confirmed symptomatic | 94 | 49 | 85
  Severe or BG confirmed | 119 | 66 | 105
  Unclassifiable | 137 | 100 | 109

49. Secondary Outcome: Number of Treatment Emergent Meal Related (From Start of Meal Until 2 Hours After Start of Meal) Hypoglycaemic Episodes According to Novo Nordisk/ISPAD Classification
Description: as for outcome 48
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 2 | 1 | 1
  BG confirmed | 715 | 504 | 600
  Severe or BG confirmed symptomatic | 572 | 414 | 495
  Severe or BG confirmed | 717 | 505 | 601
  Unclassifiable | 838 | 653 | 730

50. Secondary Outcome: Number of Treatment Emergent Meal Related (From Start of Meal Until 4 Hours After Start of Meal) Hypoglycaemic Episodes According to Novo Nordisk/ISPAD Classification
Description: as for outcome 48
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 3 | 1 | 2
  BG confirmed | 1774 | 1781 | 1666
  Severe or BG confirmed symptomatic | 1365 | 1375 | 1277
  Severe or BG confirmed | 1777 | 1782 | 1668
  Unclassifiable | 2628 | 2503 | 2347

51. Secondary Outcome: Number of Treatment Emergent Meal Related (From 2-4 Hours After Start of Meal) Hypoglycaemic Episodes According to Novo Nordisk/ISPAD Classification
Description: as for outcome 48
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Episodes
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Episodes
  Severe | 1 | 0 | 1
  BG confirmed | 1059 | 1277 | 1066
  Severe or BG confirmed symptomatic | 793 | 961 | 782
  Severe or BG confirmed | 1060 | 1277 | 1067
  Unclassifiable | 1790 | 1850 | 1617

52. Secondary Outcome: Number of Treatment Emergent Adverse Events (AEs)
Description: Treatment emergent was defined as an event that has onset up to 7 days after last day of IMP (faster aspart or NovoRapid®/NovoLog®) and excluding the events occurring in the run-in period. The results are based on the on-treatment period.
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Events
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Events | 576 | 678 | 593

53. Secondary Outcome: Number of Treatment Emergent Injection Site Reactions
Description: Treatment emergent was defined as an event that has onset up to 7 days after last day of IMP and excluding the events occurring in the run-in period. The results are based on the on-treatment period.
Time Frame: Week 0-26
Population: as for outcome 12
Measure: Number; unit: Events
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Events | 11 | 31 | 17

54. Secondary Outcome: Change in Physical Examination
Description: The following physical examinations were done: 1) Cardiovascular system. 2) Central and peripheral nervous system. 3) Gastrointestinal system including the mouth. 4) General appearance. 5) Head, ears, eyes, nose, throat and neck. 6) Musculoskeletal system. 7) Respiratory system. 8) Skin. Presented results are number of participants with the following outcomes: normal, abnormal not clinically significant (NCS) and abnormal clinically significant (CS). Presented results are baseline (week 0) and last on-treatment values. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Participants
  1) Baseline: Normal | 260 | 254 | 258
  1) Baseline: Abnormal, NCS | 1 | 4 | 0
  1) Baseline: Abnormal, CS | 0 | 0 | 0
  1) Last on-treatment: Normal: number analyzed (Participants) | 257 | 258 | 257
  1) Last on-treatment: Normal | 257 | 253 | 257
  1) Last on-treatment: Abnormal, NCS: number analyzed (Participants) | 257 | 258 | 257
  1) Last on-treatment: Abnormal, NCS | 0 | 5 | 0
  1) Last on-treatment: Abnormal, CS: number analyzed (Participants) | 257 | 258 | 257
  1) Last on-treatment: Abnormal, CS | 0 | 0 | 0
  2) Baseline: Normal | 257 | 253 | 258
  2) Baseline: Abnormal, NCS | 3 | 4 | 0
  2) Baseline: Abnormal, CS | 1 | 1 | 0
  2) Last on-treatment: Normal: number analyzed (Participants) | 257 | 258 | 257
  2) Last on-treatment: Normal | 255 | 253 | 257
  2) Last on-treatment: Abnormal, NCS: number analyzed (Participants) | 257 | 258 | 257
  2) Last on-treatment: Abnormal, NCS | 2 | 4 | 0
  2) Last on-treatment: Abnormal, CS: number analyzed (Participants) | 257 | 258 | 257
  2) Last on-treatment: Abnormal, CS | 0 | 1 | 0
  3) Baseline: Normal | 258 | 257 | 254
  3) Baseline: Abnormal, NCS | 3 | 1 | 3
  3) Baseline: Abnormal, CS | 0 | 0 | 1
  3) Last on-treatment: Normal: number analyzed (Participants) | 257 | 258 | 257
  3) Last on-treatment: Normal | 253 | 257 | 256
  3) Last on-treatment: Abnormal, NCS: number analyzed (Participants) | 257 | 258 | 257
  3) Last on-treatment: Abnormal, NCS | 4 | 1 | 0
  3) Last on-treatment: Abnormal, CS: number analyzed (Participants) | 257 | 258 | 257
  3) Last on-treatment: Abnormal, CS | 0 | 0 | 1
  4) Baseline: Normal | 258 | 253 | 254
  4) Baseline: Abnormal, NCS | 2 | 3 | 4
  4) Baseline: Abnormal, CS | 1 | 2 | 0
  4) Last on-treatment: Normal: number analyzed (Participants) | 257 | 258 | 257
  4) Last on-treatment: Normal | 257 | 253 | 254
  4) Last on-treatment: Abnormal, NCS: number analyzed (Participants) | 257 | 258 | 257
  4) Last on-treatment: Abnormal, NCS | 0 | 4 | 3
  4) Last on-treatment: Abnormal, CS: number analyzed (Participants) | 257 | 258 | 257
  4) Last on-treatment: Abnormal, CS | 0 | 1 | 0
  5) Baseline: Normal | 251 | 238 | 245
  5) Baseline: Abnormal, NCS | 9 | 13 | 11
  5) Baseline: Abnormal, CS | 1 | 7 | 2
  5) Last on-treatment: Normal: number analyzed (Participants) | 257 | 258 | 257
  5) Last on-treatment: Normal | 247 | 244 | 242
  5) Last on-treatment: Abnormal, NCS: number analyzed (Participants) | 257 | 258 | 257
  5) Last on-treatment: Abnormal, NCS | 7 | 11 | 14
  5) Last on-treatment: Abnormal, CS: number analyzed (Participants) | 257 | 258 | 257
  5) Last on-treatment: Abnormal, CS | 3 | 3 | 1
  6) Baseline: Normal | 259 | 252 | 254
  6) Baseline: Abnormal, NCS | 2 | 4 | 3
  6) Baseline: Abnormal, CS | 0 | 2 | 1
  6) Last on-treatment: Normal: number analyzed (Participants) | 257 | 258 | 257
  6) Last on-treatment: Normal | 254 | 253 | 253
  6) Last on-treatment: Abnormal, NCS: number analyzed (Participants) | 257 | 258 | 257
  6) Last on-treatment: Abnormal, NCS | 1 | 3 | 3
  6) Last on-treatment: Abnormal, CS: number analyzed (Participants) | 257 | 258 | 257
  6) Last on-treatment: Abnormal, CS | 2 | 2 | 1
  7) Baseline: Normal | 259 | 256 | 256
  7) Baseline: Abnormal, NCS | 1 | 2 | 1
  7) Baseline: Abnormal, CS | 1 | 0 | 1
  7) Last on-treatment: Normal: number analyzed (Participants) | 257 | 258 | 257
  7) Last on-treatment: Normal | 257 | 258 | 257
  7) Last on-treatment: Abnormal, NCS: number analyzed (Participants) | 257 | 258 | 257
  7) Last on-treatment: Abnormal, NCS | 0 | 0 | 0
  7) Last on-treatment: Abnormal, CS: number analyzed (Participants) | 257 | 258 | 257
  7) Last on-treatment: Abnormal, CS | 0 | 0 | 0
  8) Baseline: Normal | 239 | 237 | 238
  8) Baseline: Abnormal, NCS | 18 | 21 | 16
  8) Baseline: Abnormal, CS | 4 | 0 | 4
  8) Last on-treatment: Normal: number analyzed (Participants) | 257 | 258 | 257
  8) Last on-treatment: Normal | 229 | 233 | 235
  8) Last on-treatment: Abnormal, NCS: number analyzed (Participants) | 257 | 258 | 257
  8) Last on-treatment: Abnormal, NCS | 19 | 22 | 17
  8) Last on-treatment: Abnormal, CS: number analyzed (Participants) | 257 | 258 | 257
  8) Last on-treatment: Abnormal, CS | 9 | 3 | 5

55. Secondary Outcome: Change in Vital Sign: Blood Pressure
Description: Change from baseline (week 0) in blood pressure (systolic blood pressure (SBP) and diastolic blood pressure (DBP)) was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value.
Time Frame: Week 0, Week 26
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmHg
  SBP: Baseline | 106.4 (11.8) | 107.0 (12.6) | 106.8 (11.4)
  SBP: Change from baseline | 0.8 (11.0) | 1.5 (10.4) | 1.1 (10.1)
  DBP: Baseline | 65.4 (8.3) | 65.7 (9.4) | 65.4 (7.9)
  DBP: Change from baseline | 1.2 (9.1) | 1.4 (9.3) | 1.4 (8.3)

56. Secondary Outcome: Change in Vital Sign: Pulse
Description: Change from baseline (week 0) in pulse was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value.
Time Frame: Week 0, Week 26
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Beats/minute
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Beats/minute
  Baseline | 80.6 (11.8) | 80.5 (11.8) | 79.4 (11.8)
  Change from baseline | -0.6 (10.3) | 0.3 (10.8) | 0.7 (11.0)

57. Secondary Outcome: Change in Body Weight
Description: Change from baseline (week 0) in body weight was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: SAS. One participant was randomised to the postmeal faster aspart group but was exposed to mealtime faster aspart throughout the study. The participant was included in the mealtime faster aspart group for the SAS. Therefore, number of participants analysed at baseline= Faster aspart (meal): 261, Faster aspart (post): 258 and NovoRapid (meal): 258.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
kg
  Baseline | 46.69 (18.15) | 46.48 (18.98) | 46.28 (17.18)
  Change from baseline: number analyzed (Participants) | 257 | 258 | 257
  Change from baseline | 2.21 (2.57) | 1.90 (2.32) | 2.15 (2.80)

58. Secondary Outcome: Change in Height
Description: Change from baseline (week 0) in height was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: Meter
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Meter
  Baseline | 1.50 (0.21) | 1.50 (0.21) | 1.50 (0.19)
  Change from baseline: number analyzed (Participants) | 257 | 258 | 257
  Change from baseline | 0.02 (0.02) | 0.02 (0.02) | 0.02 (0.02)

59. Secondary Outcome: Change in Body Mass Index
Description: Change from baseline (week 0) in body mass index (BMI) was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
kg/m^2
  Baseline: number analyzed (Participants) | 260 | 258 | 258
  Baseline | 19.68 (3.75) | 19.67 (4.02) | 19.64 (3.78)
  Change from baseline: number analyzed (Participants) | 257 | 258 | 257
  Change from baseline | 0.37 (0.92) | 0.28 (0.92) | 0.34 (1.10)

60. Secondary Outcome: Change in SD Score of Body Weight
Description: Change from baseline (week 0) in standard deviation (SD) score of body weight was evaluated after 26 weeks of randomisation. SD-scores are defined to be able to normalise the body weight in the various age groups. To estimate the growth of children, standardised weight is calculated for each year of age and for each sex. Thus, a child with a weight equal to the mean value for its age and sex has an SD score of 0, while a child with a weight 2 SDs above the mean value for its age and sex has an SD score of +2. The SD scores are derived from the age and sex of the subjects and the body weight together with growth curves defined for a reference population. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Standard deviation score
  Baseline: number analyzed (Participants) | 260 | 258 | 258
  Baseline | 0.349 (0.945) | 0.351 (0.936) | 0.361 (0.875)
  Change from baseline: number analyzed (Participants) | 257 | 258 | 257
  Change from baseline | 0.034 (0.231) | 0.008 (0.223) | 0.030 (0.250)

61. Secondary Outcome: Change in SD Score of Body Mass Index
Description: Change from baseline (week 0) in SD score of BMI was evaluated after 26 weeks of randomisation. SD scores for BMI were determined in a similar way as SD scores for weight by use of a suitable reference population based on age and sex. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: Standard deviation score
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Standard deviation score
  Baseline: number analyzed (Participants) | 260 | 258 | 258
  Baseline | 0.296 (0.895) | 0.298 (0.936) | 0.317 (0.898)
  Change from baseline: number analyzed (Participants) | 257 | 258 | 257
  Change from baseline | 0.016 (0.308) | 0.004 (0.370) | 0.007 (0.338)

62. Secondary Outcome: Change in Haematology: Haemoglobin
Description: Change from baseline (week 0) in haemoglobin was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline | 8.33 (0.72) | 8.47 (0.74) | 8.41 (0.77)
  Change from baseline: number analyzed (Participants) | 257 | 258 | 257
  Change from baseline | 0.08 (0.51) | 0.09 (0.62) | 0.09 (0.52)

63. Secondary Outcome: Change in Haematology: Haematocrit
Description: Change from baseline (week 0) in haematocrit was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: % of red blood cells
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
% of red blood cells
  Baseline | 40.87 (3.39) | 41.51 (3.50) | 41.34 (3.75)
  Change from baseline: number analyzed (Participants) | 257 | 257 | 257
  Change from baseline | 0.45 (2.86) | 0.40 (3.09) | 0.32 (2.75)

64. Secondary Outcome: Change in Haematology: Erythrocytes
Description: Change from baseline (week 0) in erythrocytes was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
10^12 cells/L
  Baseline | 4.81 (0.39) | 4.87 (0.39) | 4.88 (0.40)
  Change from baseline: number analyzed (Participants) | 257 | 258 | 257
  Change from baseline | 0.02 (0.27) | 0.04 (0.31) | 0.02 (0.26)

65. Secondary Outcome: Change in Haematology: Thrombocytes
Description: Change from baseline (week 0) in thrombocytes was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
10^9 cells/L
  Baseline | 268.1 (64.5) | 270.0 (60.2) | 262.5 (57.9)
  Change from baseline: number analyzed (Participants) | 257 | 258 | 257
  Change from baseline | 1.2 (47.3) | 1.6 (45.4) | 6.0 (44.9)

66. Secondary Outcome: Change in Haematology: Leukocytes
Description: Change from baseline (week 0) in leukocytes was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
10^9 cells/L
  Baseline | 6.10 (1.65) | 6.10 (1.63) | 6.11 (1.81)
  Change from baseline: number analyzed (Participants) | 257 | 258 | 257
  Change from baseline | 0.08 (1.66) | 0.14 (1.74) | 0.10 (1.67)

67. Secondary Outcome: Change in Biochemistry: Creatinine
Description: Change from baseline (week 0) in creatinine was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
umol/L
  Baseline | 51.8 (14.2) | 52.6 (13.3) | 52.1 (12.3)
  Change from baseline: number analyzed (Participants) | 257 | 257 | 256
  Change from baseline | 1.1 (7.8) | 1.5 (6.9) | 1.7 (6.8)

68. Secondary Outcome: Change in Biochemistry: Alanine Aminotransferase (ALT)
Description: Change from baseline (week 0) in ALT was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
U/L
  Baseline | 14.4 (6.4) | 14.7 (7.4) | 14.8 (5.6)
  Change from baseline: number analyzed (Participants) | 257 | 257 | 256
  Change from baseline | 0.1 (6.9) | 1.3 (14.9) | 0.5 (5.9)

69. Secondary Outcome: Change in Biochemistry: Aspartate Aminotransferase (AST)
Description: Change from baseline (week 0) in AST was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
U/L
  Baseline | 19.9 (6.8) | 20.0 (5.6) | 20.5 (5.9)
  Change from baseline: number analyzed (Participants) | 257 | 257 | 256
  Change from baseline | 0.1 (6.2) | 1.1 (11.7) | -0.4 (5.0)

70. Secondary Outcome: Change in Biochemistry: Alkaline Phosphatase (AP)
Description: Change from baseline (week 0) in AP was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
U/L
  Baseline | 212.7 (135.8) | 209.8 (94.9) | 226.2 (93.6)
  Change from baseline: number analyzed (Participants) | 257 | 257 | 256
  Change from baseline | -3.0 (119.0) | -1.7 (50.8) | -2.8 (80.4)

71. Secondary Outcome: Change in Biochemistry: Sodium
Description: Change from baseline (week 0) in sodium was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline | 139.5 (2.5) | 139.6 (2.4) | 139.7 (2.5)
  Change from baseline: number analyzed (Participants) | 257 | 257 | 256
  Change from baseline | 0.5 (2.8) | 0.3 (2.7) | 0.04 (2.8)

72. Secondary Outcome: Change in Biochemistry: Potassium
Description: Change from baseline (week 0) in potassium was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
mmol/L
  Baseline | 4.48 (0.34) | 4.52 (0.34) | 4.52 (0.40)
  Change from baseline: number analyzed (Participants) | 257 | 257 | 256
  Change from baseline | 0.02 (0.41) | -0.06 (0.34) | 0.01 (0.50)

73. Secondary Outcome: Change in Biochemistry: Albumin
Description: Change from baseline (week 0) in albumin was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
g/dL
  Baseline | 4.47 (0.24) | 4.51 (0.24) | 4.50 (0.25)
  Change from baseline: number analyzed (Participants) | 257 | 257 | 256
  Change from baseline | 0.01 (0.24) | 0.01 (0.25) | 0.005 (0.24)

74. Secondary Outcome: Change in Biochemistry: Total Bilirubin
Description: Change from baseline (week 0) in total bilirubin was evaluated after 26 weeks of randomisation. The results are based on the last on-treatment value. Number of participants analysed = number of participants contributed to the analysis.
Time Frame: Week 0, Week 26
Population: as for outcome 57
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
umol/L
  Baseline | 7.9 (6.0) | 7.9 (5.3) | 8.0 (6.2)
  Change from baseline: number analyzed (Participants) | 257 | 256 | 256
  Change from baseline | 0.2 (4.9) | 0.2 (3.4) | 0.3 (4.1)

75. Secondary Outcome: Change in Lipid Profile: Total Cholesterol
Description: Change from baseline (week 0) in total cholesterol after 26 weeks of randomisation is presented as ratio to baseline values. The results are based on the last on-treatment value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Ratio | 0.989 (13.869) | 1.023 (13.742) | 1.016 (13.187)

76. Secondary Outcome: Change in Lipid Profile: High Density Lipoproteins (HDL)
Description: Change from baseline (week 0) in HDL after 26 weeks of randomisation is presented as ratio to baseline values. The results are based on the last on-treatment value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Ratio | 1.004 (17.865) | 1.030 (20.180) | 1.023 (17.852)

77. Secondary Outcome: Change in Lipid Profile: Low Density Lipoproteins (LDL)
Description: Change from baseline (week 0) in LDL after 26 weeks of randomisation is presented as ratio to baseline values. The results are based on the last on-treatment value.
Time Frame: Week 0, Week 26
Population: FAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Ratio | 1.014 (19.533) | 1.040 (19.685) | 1.041 (19.864)

78. Secondary Outcome: Change in Anti-insulin Aspart Antibody Development: Specific
Description: Change from baseline (week 0) in 'antibodies specific for insulin aspart' was evaluated after 26 weeks of randomisation. This endpoint was measured as % bound radioactivity-labelled insulin aspart/Total added radioactivity-labelled insulin aspart (%B/T). The results are based on the last on-treatment value.
Time Frame: Week 0, Week 26
Population: SAS. One participant was randomised to the postmeal faster aspart group but was exposed to mealtime faster aspart throughout the study. The participant was included in the mealtime faster aspart group for the SAS. Number of participants analysed = number of participants contributed to the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of B/T
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Percentage of B/T
  Baseline: number analyzed (Participants) | 258 | 256 | 253
  Baseline | 1.436 (3.159) | 1.459 (5.313) | 1.183 (2.134)
  Change from baseline: number analyzed (Participants) | 254 | 256 | 252
  Change from baseline | -0.099 (1.015) | -0.213 (1.661) | -0.201 (1.238)

79. Secondary Outcome: Change in Anti-insulin Aspart Antibody Development: Cross-reacting With Human Insulin
Description: Change from baseline (week 0) in 'antibodies for insulin aspart, those cross-reacting with human insulin' was evaluated after 26 weeks of randomisation. This endpoint was measured as % bound radioactivity-labelled insulin aspart/Total added radioactivity-labelled insulin aspart (%B/T). The results are based on the last on-treatment value.
Time Frame: Week 0, Week 26
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Percentage of B/T
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Percentage of B/T
  Baseline: number analyzed (Participants) | 258 | 254 | 252
  Baseline | 18.794 (17.189) | 21.576 (17.721) | 20.156 (17.315)
  Change from baseline: number analyzed (Participants) | 254 | 254 | 251
  Change from baseline | -3.202 (6.989) | -4.845 (7.034) | -3.802 (7.587)

80. Secondary Outcome: Change in Anti-insulin Aspart Antibody Development: Total
Description: Change from baseline (week 0) in 'total anti-insulin aspart antibodies (specific for insulin aspart and those cross-reacting with human insulin)' was evaluated after 26 weeks of randomisation. This endpoint was measured as % bound radioactivity-labelled insulin aspart/Total added radioactivity-labelled insulin aspart (%B/T). The results are based on the last on-treatment value.
Time Frame: Week 0, Week 26
Population: as for outcome 78
Measure: Mean (Standard Deviation); unit: Percentage of B/T
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
Number analyzed (Participants) | 260 | 259 | 258
Percentage of B/T
  Baseline: number analyzed (Participants) | 258 | 254 | 252
  Baseline | 20.230 (17.795) | 23.044 (18.070) | 21.344 (17.825)
  Change from baseline: number analyzed (Participants) | 254 | 254 | 251
  Change from baseline | -3.271 (7.158) | -5.061 (7.193) | -4.004 (7.700)

ADVERSE EVENTS:
Time Frame: Week 0 to week 26 + 7 days. Presented adverse events are treatment emergent.
Description: SAS. One participant was randomised to the postmeal faster aspart group but was exposed to mealtime faster aspart throughout the study. The participant was included in the mealtime faster aspart group for the SAS. Therefore, number of participants analysed at baseline= Faster aspart (meal): 261, Faster aspart (post): 258 and NovoRapid (meal): 258.
Arm/Group | Faster Aspart (Meal) | Faster Aspart (Post) | NovoRapid (Meal)
All-Cause Mortality (participants affected / at risk) | 0/261 | 0/258 | 0/258
Serious Adverse Events (participants affected / at risk) | 5/261 | 13/258 | 9/258
Other Adverse Events (participants affected / at risk) | 137/261 | 149/258 | 136/258
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart (Meal) (N=261) | Faster Aspart (Post) (N=258) | NovoRapid (Meal) (N=258)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Adjustment disorder with mixed disturbance of emotion and conduct (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus management (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 2 (2)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)
Gastrointestinal viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Idiopathic partial epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart (Meal) (N=261) | Faster Aspart (Post) (N=258) | NovoRapid (Meal) (N=258)
Cough (Respiratory, thoracic and mediastinal disorders) | 10 (11) | 11 (14) | 16 (21)
Gastroenteritis (Infections and infestations) | 13 (15) | 16 (17) | 19 (24)
Headache (Nervous system disorders) | 16 (21) | 26 (38) | 22 (35)
Influenza (Infections and infestations) | 20 (28) | 14 (19) | 14 (21)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 9 (13) | 13 (16)
Pyrexia (General disorders) | 22 (26) | 16 (16) | 18 (20)
Rhinitis (Infections and infestations) | 10 (16) | 16 (24) | 11 (16)
Upper respiratory tract infection (Infections and infestations) | 22 (31) | 32 (41) | 26 (32)
Viral infection (Infections and infestations) | 7 (8) | 9 (11) | 14 (20)
Viral upper respiratory tract infection (Infections and infestations) | 60 (73) | 53 (79) | 48 (75)
Vomiting (Gastrointestinal disorders) | 9 (9) | 21 (24) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property

DOCUMENTS (2):
  • Study Protocol (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT02670915/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-17): https://cdn.clinicaltrials.gov/large-docs/15/NCT02670915/SAP_001.pdf